CLINICAL TRIAL: NCT02781688
Title: Increasing Physical Activity in Persons With Depression - Pilot
Brief Title: Increasing Physical Activity in Persons With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 092015-038
Record Dates: First submitted 2016-05-03; First posted 2016-05-24 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Depression; Physical Activity
MeSH Terms: conditions — Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical Activity Intervention (Experimental): Participants will participate in a multi-component physical activity intervention for 12 weeks.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Self-monitoring: Subjects will be provided with a commercially available activity monitor (i.e., Fitbit) and instructed to wear the device daily.
  Active Living counseling: The Active Living counseling program will consists of 12 weekly group educational sessions, facilitated by project interventionists. These sessions will involve discussion of topics related to increasing physical activity, including: identifying and overcoming barriers, setting goals, social support, and time management.
  Facility Access: Subjects will have access to the exercise lab in the UT Southwestern Depression Center consisting of equipment for aerobic exercise (treadmills, stationary bikes, etc.).

SUMMARY:
Pilot study to assess a multi-component intervention to increase physical activity in persons with depression.

DETAILED DESCRIPTION:
The research project is a pilot study to assess the effects of a multi-component intervention in increasing physical activity among persons with depression. Individuals meeting inclusion/exclusion criteria will be enrolled in the 12-week intervention. Intervention components will include self-monitoring, Active Living counseling, and facility access. Blood samples will be collected at baseline. Assessments (anxiety, stress, sleep) and sample collection will also occur at 2 time points during the intervention (Weeks 7 and 13). Changes in physical activity will be assessed using Fitbits to measure weekly minutes of moderate/vigorous activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Positive depression screen (Patient Health Questionnaire [PHQ-9]) or current antidepressant treatment
* Report <150 minutes of weekly moderate-to-vigorous physical activity (MVPA) on the Exercise Vital Sign (EVS)
* Written and verbal fluency in English

Exclusion Criteria:

* Medical condition contraindicating physical activity participation
* Cognitively unable to give informed consent
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity as measured by Actigraph accelerometer | 12 weeks
  Assess changes in minutes of moderate-to-vigorous physical activity (MVPA) at 3 months following physical activity intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No